CLINICAL TRIAL: NCT02343536
Title: A Phase 1, Open-label, Multicenter Trial of Oral Azacitidine (CC-486) Plus R-CHOP in Subjects With High Risk (IPI 3 or More) Previously Untreated Diffuse Large B-cell Lymphoma or Grade 3B Follicular Lymphoma.
Brief Title: A Phase 1, Open-label Trial of Oral Azacitidine (CC-486) Plus RCHOP in Subjects With Large B-Cell Lymphoma or Follicular Lymphoma or Transformed Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-486-DLBCL-001
Expanded Access: NCT03723135 (Approved for marketing)
Record Dates: First submitted 2015-01-16; First posted 2015-01-22 (Estimated); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular
Keywords: Phase 1; Oral Azacitidine (CC-486); R-CHOP; Diffuse Large B-cell Lymphoma; Grade 3B Follicular Lymphoma; Follicular Lymphoma; Transformed Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular | interventions — Azacitidine; cc-486; Rituximab; Cyclophosphamide; Vincristine; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oral Azacitidine (CC-486) and R-CHOP (Experimental): Will examine four escalating dose-levels of CC- 486 (100 mg, 150 mg, 200 mg and 300 mg).
  Interventions: Drug: Oral Azacitidine; Drug: Rituximab; Drug: cyclophosphamide; Drug: Vincristine; Drug: Prednisone
- R-CHOP (Active Comparator): R-CHOP, (rituximab, cyclophosphamide, doxorubicin, vincristine, prednisone) * rituximab, cyclophosphamide, doxorubicin, and vincristine are administered on Day 1; while prednisone is administered Days 1-5
  Interventions: Drug: Rituximab; Drug: cyclophosphamide; Drug: Vincristine; Drug: Prednisone

INTERVENTIONS:
Drug: Oral Azacitidine
  Other Names: CC-486
  Arms: Oral Azacitidine (CC-486) and R-CHOP
Drug: Rituximab
Drug: cyclophosphamide
Drug: Vincristine
Drug: Prednisone

SUMMARY:
The goal of the study is to identify a dose and schedule of CC-486 that can be safely administered with R-CHOP. To evaluate the safety and maximum tolerated dose (MTD) or the maximal administered dose (MAD) of CC-486 in combination with rituximab, cyclophosphamide, doxorubicin, vincristine, and prednisone (R-CHOP) in subjects with high risk (IPI 2 or more) previously untreated DLBCL or Grade 3B FL.

Also, to determine pharmacokinetics (PK) of CC-486 when administered alone and in combination with R-CHOP and to explore preliminary efficacy of CC-486 plus R-CHOP by 2007 International Working Group (IWG) criteria.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety of oral azacitidine (CC-486) when combined with R-CHOP (the treatment regimen normally used in treating Diffuse large B-cell lymphoma or Grade 3B follicular lymphoma). This study also proposes to explore the pharmacokinetics of oral azacitidine when administered in combination with R-CHOP and to assess the effects the drug can have on the human body, as well as the ability of CC 486 in combination with R CHOP to further effect the response of tumors associated with Diffuse large B-cell lymphoma or Grade 3B follicular lymphoma, .

Oral azacitidine in combination with R-CHOP has not been approved for the treatment of Diffuse large B-cell lymphoma or Grade 3B follicular lymphoma and its use in this study is investigational. Various dose levels of this investigation treatment will be administered to subject enrolled into the study.

This study is separated into three periods: Screening and Registration, Treatment and Follow-up periods. Before the patient can receive the study drug the doctor will perform tests to find out whether he/she can participate in the study. This is done during the Screening Period. If the patient and the treating physician determine that the patient is eligible to participate in the study, the patient will be registered in the study and assigned to receive one of the investigational dose levels of oral azacitidine.

The Treatment period starts when the patient receives their first dose of the study drug. The maximum time the patient will receive study treatment is 5 months. The intent is for the patient to complete 6 cycles of treatment. Each cycle will be 21 days. The Follow-up period starts when the patient's treatment is completed or discontinued for any reason. The patient will have fewer exams, tests and visits once entering the follow-up period. These visits will be every 6 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed previously untreated DLBCL or Grade 3B FL, [double-positive for BCL2 and c-MYC] or transformed lymphoma. Transformed lymphoma from FL or marginal zone lymphoma, but not chronic lymphocytic leukemia (CLL) [Richter Transformation] are allowed as long as no prior anti-lymphoma therapy of any kind has been administered.

   1. A formalin fixed paraffin embedded lymph node or tumor biopsy specimen must be submitted during the Screening Period. The specimen must have been acquired by a surgical or core needle biopsy (≥ 2 cores at baseline); material from a fine needle aspiration is not acceptable.
   2. Fresh core biopsy, frozen, must be performed before start of therapy and submitted for storage. This is optional only for the subjects who have a biopsy-accessible site and consent to the procedure. In case no prior fixed formalin paraffin embedded (FFPE) biopsy is available, this specimen can also be used for diagnostic confirmation.
   3. No prior anti-lymphoma therapy. However, for subjects with bulky disease,systemic symptoms, compressive disease, or rapidly progressing adenopathies, pre-phase treatment with 1 mg/kg/day prednisone, or equivalent, for a maximum of 7 days is permitted prior to Cycle 1 Day -6 at the discretion of the Investigator. In exceptional cases, if clinically indicated, a higher dose of steroids and/or a slightly longer duration is allowed for the purpose of urgent symptom management, and the subjects is considered eligible. A washout period does not apply. However the fresh core biopsy mentioned above should be performed before starting prednisone.
2. International Prognostic Index score ≥ 2 or DLBCL with double-positive for BCL2 and c-MYC by IHC (immunohistochemistry) or FISH (fluorescent in situ hybridization) based on local pathology lab assessment.
3. Measurable disease on cross section imaging by CT (computed tomography) that is at least 1.5 cm in the longest diameter and measurable in two perpendicular dimensions as defined by IWG (International Working Group) response criteria for NHL (non-Hodgkin Lymphoma).
4. Ann Arbor stage II to IV.
5. Men and women 18 years of age to 80 years of age of any ethnic origin or race at the time of signing the ICD.
6. Understand and voluntarily sign an ICD (Informed Consent Document) prior to any study related assessments/procedures are conducted.
7. Able to adhere to the study visit schedule and other protocol requirements.
8. Performance status ≤ 2 on the Eastern Cooperative Oncology Group (ECOG) scale.
9. Negative serum pregnancy test within 72 hours before starting study treatment on Cycle 1 Day -6 for females of childbearing potential (FCBP). A female of child-bearing potential, defined as a sexually mature woman who: 1) has not undergone a hysterectomy (the surgical removal of the uterus) or bilateral oophorectomy (the surgical removal of both ovaries) or, 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time during the preceding 24 consecutive months), may participate providing they agree to the following conditions:

   1. Either commit to true abstinence* from heterosexual contact (which must be reviewed on a monthly basis) or agree to the use of a physician-approved contraceptive method (oral, injectable, or implantable hormonal contraceptive; tubal ligation; intrauterine device; barrier contraceptive with spermicide; or vasectomized partner) without interruption, while on CC-486 (including dose interruptions); and for 3 months following the last dose of IP; and
   2. Agree to have a medically supervised serum pregnancy test with sensitivity of at least 25 mIU/mL obtained at Screening. A serum pregnancy test is to be performed within 72 hours prior to Day 1 of starting study therapy on Cycle 1 Day -6, and within 72 hours prior to Day 1 of every subsequent cycle, and at the Treatment Discontinuation Visit. The subject may not receive IP until the Investigator has verified that the result of the pregnancy test is negative.
10. Male subjects with a female partner of childbearing potential must either commit to true abstinence* or agree to the use of a physician-approved contraceptive method throughout the course of the study and avoid fathering a child during the course of the study and for 3 months following the last dose of the IP (Investigational Product).

Exclusion Criteria:

1. Any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study.
2. Any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study.
3. Any condition that confounds the ability to interpret data from the study.
4. Any condition causing an inability to swallow tablets.
5. History of inflammatory bowel disease (e.g., Crohnis disease, ulcerative colitis),celiac disease (i.e., sprue), prior gastrectomy or upper bowel removal, or any other gastrointestinal disorder or defect that would interfere with absorption, distribution, metabolism, or excretion of the IP and/or predispose the subject to an increased risk of gastrointestinal toxicity.
6. Hematologic and Non-hematologic exclusion criteria before start of therapy.
7. Seropositive for or active viral infection with hepatitis B virus (HBV):

   1. Hepatitis B surface antigen (HBsAg) positive
   2. HBsAg negative, anti-HBs positive and/or anti-HBc positive and detectable viral DNA
   3. Subjects who are HBsAg negative, anti-HBs positive, and/or anti-HBc positive, but viral DNA negative are not eligible
   4. Subjects who are seropositive because of HBV vaccination are eligible (HBV surface antibody positive, HBV core antibody negative, and HBV surface antigen negative)
8. Prior history of malignancies, other than diffuse large B-cell lymphoma, unless the subject has been free of the disease for ≥ 5 years from the signing of the ICD. Exceptions to the ≥ 5 year time limit include history of the following:

   1. Basal cell carcinoma of the skin
   2. Squamous cell carcinoma of the skin
   3. Carcinoma in situ of the cervix
   4. Carcinoma in situ of the breast
   5. Incidental histological finding of prostate cancer (TNM stage of T1a or T1b)
9. Known seropositive for or active infection with hepatitis C virus (HCV)
10. Known seropositive for or active viral infection with human immunodeficiency virus (HIV).
11. Known or suspected hypersensitivity to azacitidine or mannitol or any other ingredient used in the manufacture of oral azacitidine (see the current azacitidine IB).
12. Contraindication to any drug in the chemotherapy regimen, and specifically

    1. LVEF < 50%
    2. Corrected QT interval > 480 msec (using the Fridericia formula)
    3. Neuropathy uropathy europathy Nemediastinal DLBCL.
13. Primary mediastinal DLBCL.
14. Active uncontrolled systemic fungal, bacterial, or viral infection (defined as ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics, antiviral therapy, and/or other treatment)
15. Significant active cardiac disease within the previous 6 months from the signing of the ICD, including:

    1. New York Heart Association (NYHA) class III or IV congestive heart failure
    2. Unstable angina or angina requiring surgical or medical intervention; and/or
    3. Myocardial infarction
16. Pregnant or lactating (breastfeeding) females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2015-04-29 (Actual); Primary Completion 2020-01-29 (Actual); Study Completion 2020-01-29 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 1 year
  The dose level corresponding to the target Dose Limiting Toxicity (DLT) probability of 0.20.
Maximal Administered Dose (MAD) | 1 Year
  The highest recorded dose administered to a subject if the MTD is not reached
Adverse Event (AE) | 2 Years
  Number of participants with adverse events

SECONDARY OUTCOMES:
Pharmacokinetics- Cmax | 2 Years
  Maximum observed concentration in plasma
Pharmacokinetics - AUC | 2 Years
  Area under the concentration-time curve
Pharmacokinetics - Tmax | 2 Years
  Time to maximum concentration
Pharmacokinetics - t1/2 | 2 Years
  Terminal half-life
Pharmacokinetics CL/F | 2 Years
  Apparent total body clearance
Pharmacokinetics - Vz/F | 2 Years
  Apparent volume of distribution
Overall response rate (ORR) | 4 Years
  Efficacy evaluation of CC-486 plus R-CHOP of the percentage of subjects achieving and clinical response (Complete or Partial Remission) as assessed by 2007 International Working Group (IWG) criteria for non-Hodgkin lymphoma as evaluated by investigator review.
Complete response (CR) rate | 4 Years
  Efficacy evaluation of CC-486 plus R-CHOP of the percentage of subjects achieving Complete Remission as assessed by 2007 International Working Group (IWG) criteria for non-Hodgkin lymphoma as evaluated by investigator review.
Progression free survival (PFS) | 4 Years
  Efficacy evaluation of CC-486 plus R-CHOP. Progression-free survival is calculated as the time from C1D1 to the first documented progression or death due to any cause. Progression will be assessed by 2007 International Working Group (IWG) criteria for non-Hodgkin lymphoma as evaluated by investigator review.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zhang, MD, Study Director — Celgene
Locations (7):
- United States (7):
  - Moffitt Cancer Center, Tampa, Florida
  - University of Chicago, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Weill Cornell Medicine, New York, New York
  - Rhode Island Hospital, Providence, Rhode Island

REFERENCES:
- [Derived] Martin P, Bartlett NL, Chavez JC, Reagan JL, Smith SM, LaCasce AS, Jones J, Drew J, Wu C, Mulvey E, Revuelta MV, Cerchietti L, Leonard JP. Phase 1 study of oral azacitidine (CC-486) plus R-CHOP in previously untreated intermediate- to high-risk DLBCL. Blood. 2022 Feb 24;139(8):1147-1159. doi: 10.1182/blood.2021011679. PMID 34428285